CLINICAL TRIAL: NCT02654392
Title: Effect of Plant Omega-3 and Omega-6 Fatty Acids on Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor & Weider Research Chair Director, Exercise Nutrition Research Laboratory, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 10010467
Record Dates: First submitted 2016-01-09; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Effect of Essential Fatty Acids on Exercise Performance
Keywords: Omega-3; Omega-6; Exercise Performance
MeSH Terms: interventions — High Fructose Corn Syrup; Fatty Acids, Unsaturated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): This group will receive isoenergetic carbohydrate (corn syrup) supplement daily for 5 weeks
  Interventions: Dietary Supplement: corn syrup
- Polyunsaturated fatty acid group (Other): This group will receive a plant essential fatty acid food supplement, Pureform Omega® capsules made from Fax, Sunflower, Coconut, Evening Primrose, & Pumpkin oils, containing a 2.5:1 omega-6 to omega-3 ratio (1.5 g per 70kg body mass plus an additional 0.5 g on exercise days)
  Interventions: Dietary Supplement: Polyunsaturated fatty acid

INTERVENTIONS:
Dietary Supplement: corn syrup — This group will receive an iso-energetic corn syrup supplement everyday for 5 weeks
  Arms: placebo
Dietary Supplement: Polyunsaturated fatty acid — This groups will receive 4 capsules/70kg body mass (Pureform Omega® capsules made from Fax, Sunflower, Coconut, Evening Primrose, & Pumpkin oils) every day for 5 weeks
  Arms: Polyunsaturated fatty acid group

SUMMARY:
Many studies in the past three decades have examined the beneficial effects of omega-3 polyunsaturated fatty acids in diet and supplementation. The effect of polyunsaturated fatty acids, specifically omega-3 and omega-6, on health have been well-studied but most of the study to date has been on animal not plant sources and much less is know about their effects on exercise performance. Additionally, while positive effects have been detected for sedentary populations or those that are at risk, well-trained athletes generally have not had established advantages in taking supplements for omega-3 and omega-6 oils. There is evidence that a specific ratio of omega-6 to omega-3 is most beneficial for the human body with regards to cardiovascular and mental health. In this study, participants randomized to either a plant supplement group (pureform omega; containing Flax, Evening Primrose, Sunflower, Coconut & Pumpkin oils; Natural Product Number = 80050660) or placebo (isoenergetic sugar pills) will be subjected to both a time trial and a high intensity interval bout, where their performance and power output will be analyzed. Blood lactate and glucose concentration, as well as oxygen consumption and carbon dioxide production will also be examined to determine if there is a change in on fat oxidation after supplementation.

DETAILED DESCRIPTION:
Double-blind placebo controlled study with two groups: a PUFA supplemented group (over 5 weeks) and a placebo (corn syrup) group. Participants are matched for initial exercise performance and assigned to each of the two groups systematically so the initial group means are similar. This is done by ranking all individuals from highest to lowest and assigning the participant with the highest score randomly to the treatment group and the other to the placebo group. Then, for the next two individuals in ranking, the highest of the two is assigned to the placebo group and the other to the treatment group. This procedure is repeated for all participant pairs. Of course, this is done separately for men and women because on average the men have greater exercise performance scores.

Dosage is 3.8 capsules/70kg body mass (rounded to the nearest capsule; 1 capsule contains 369mg PUFA from Flax, Evening Primrose, Pumpkin, Sunflower, and Coconut oil; <4 Calories) or isoenergetic placebo capsules (containing corn syrup) plus 2 capsules 20 minutes prior to exercise workouts. Eighteen recreationally active student volunteers (18-35 years old) will be recruited to complete 4 exercise tests: a cycle time trial (~15 minutes), a cycle maximal power test (30 second Wingate test), a maximal aerobic power test (running treadmill test) plus a strength/endurance test (number of bench presses with 60 kg load) pre- and post 5 weeks of daily supplementation. There will an accommodation day pre-study where each participant is familiarized with the tests to be used. Each exercise test will be completed on a separate day with at least 48 hours between each test day due to the fatiguing nature of the testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* Recreationally active (defined as those who attend a gym or play sports about 2-3 times a week),
* Non-pregnant student volunteers.

Exclusion Criteria:

* Participants cannot have taken omega-3 or other polyunsaturated fatty acid supplements or undergone any systematic exercise training in the past 3 months,
* Have symptoms or take medication for respiratory, cardiovascular, metabolic, or neuromuscular disease
* Injury limiting exercise ability
* Use heart rate or blood pressure medications
* Use any medications that have side effects for dizziness, lack of motor control, or slowed reaction time
* Smoker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
change in cycle ergometer time trial | at baseline and 5 weeks after supplementation
  A 40 Km time trial test on a cycle ergometer will be conducted before and after a 5-week supplementation period
change in Aerobic capacity (VO2 max) test | at baseline and 5 weeks after supplementation
  Aerobic capacity will be quantified using an incremental running test on a treadmill. The workload will be increased by increasing the slope (simulating a hill) at a constant speed (6mph)
Change in Wingate Anaerobic Test | at baseline and 5 weeks after supplementation
  A 30 second intense effort on a cycle ergometer against a load equal to 9% of body mass. Peak power, mean power, total work and fatigue index will be recorded at the end of each sprint.
change in Strength/Endurance test | at baseline and 5 weeks after supplementation
  Number of bench presses completed (rounded to the nearest 1/2 lift) with a 60 kg load and a metromone for pacing control (30 lifts per minute) will be used and rating of perceived exertion (RPE) will be assessed immediately before and immediately after each exercise test using the Borg Scale (analog scale with verbal identifiers)

SECONDARY OUTCOMES:
change in Body composition | at baseline and 5 weeks after supplementation
  Body composition will be measured by densitometry using air displacement plethysmography with a BodPod® (involves sitting comfortably in a chamber for about 2 minutes while the space the body takes up is measured) for the measurement of fat and fat-free mass
change in Blood lactate | at baseline and 5 weeks after supplementation
  Capillary blood samples (0.6 microlitres) will be collected before and after each exercise session under standard sterile condition via standard skin prick technique for the measurement of blood lactate content using a blood lactate analyzer (Lactate Scout+).
change in Blood glucose | at baseline and 5 weeks after supplementation
  Capillary blood samples (0.6 microlitres) will be collected before and after each exercise session under standard sterile condition via standard skin prick technique for the measurement of blood glucose content using a blood glucose analyzer (Free Style Lite)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Research Laboratory, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No